CLINICAL TRIAL: NCT02558062
Title: Exploratory Clinical Study of Intrapulmonary Microdosing of the BACterial Detection Probe (BAC ONE) in Ventilator Associated Pneumonia
Brief Title: Microdosing of BAC ONE to the Distal Lung
Acronym: BAC ONE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BAC ONE
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Respiratory Infections
Keywords: Ventilator Associated Pneumonia; Distal lung
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAC ONE administration (Experimental): All participants in this clinical study will be dosed on one occasion with BAC ONE. The final dosage will be 80 µg (± 25%).
  Interventions: Other: BAC ONE administration

INTERVENTIONS:
Other: BAC ONE administration — BAC ONE will be administered to each patient during a bronchoscopy procedure. Fibre-based endomicroscopy and Cellvizio viewer software will be used to detect BAC ONE signal in the distal lung.
  Other Names: BAC ONE

SUMMARY:
Critically ill patients are often ventilated in dedicated critical care units to provide respiratory support. Despite best practice patients can often develop a condition called adult respiratory distress syndrome (ARDS), which is characterised by deterioration in their respiratory function, and changes on chest x-ray. The correct management for ARDS is identifying the underlying condition causing the deterioration and identifying appropriate targeted therapy. One such cause is pneumonia, caused by a bacterial infection in the lungs of a ventilated patient. The patients may have been ventilated due to pneumonia but they may also develop pneumonia whilst ventilated. Ventilator associated pneumonia (VAP) has significant mortality.

Despite all the clinical and laboratory data at the investigators' disposal there remains great difficulty in the accurate diagnosis of pneumonia and therefore treatment is often given empirically. Therefore, there is an urgent clinical need for accurate methods to diagnose the presence of bacteria deep in the lung in ventilated critically ill patients. As such, the investigating team have developed and synthesised an imaging agent called BAC ONE. BAC ONE will be instilled directly into the lungs of 12 patients (with and without lung infection) to assess whether it can label bacteria in the human lung.

DETAILED DESCRIPTION:
The primary objective of this study is to deliver a BAC ONE microdose to ventilated controls and patients with lung infection to assess the imaging parameters of BAC ONE over human autofluorescence and to assess if bacteria can be detected in vivo in situ within the distal lung.

The primary endpoint is to visualise the delivery of a microdose of BAC ONE and assess imaging parameters in:

* 3 mechanically ventilated patients to provide a control population (cohort 1)
* 6 bronchiectasis patients with predominant colonisation with gram-negative bacteria (cohort 2)
* 6 bronchiectasis patients with predominant colonisation with gram-positive bacteria (cohort 3)
* 3 patients with suspected pneumonia and pulmonary infiltrates in ICU (cohort 4)

For all cohorts, eligibility will be verified by a clinical trial physician after written informed consent has been obtained. For all cohorts, a bronchoscopy with lavage will be performed to harvest broncho-alveolar lavage fluid (BALF). Fibre-based endomicroscopy (FE) will be performed on up to three areas and up to 80μg (± 25%) in total of BAC ONE will be instilled in up to 3 sites.

Participants will be asked to provide additional blood and urine samples with the intention of examining for systemic uptake of the BAC ONE probe. Routine blood investigations will be performed 4-6 hours following the administration of BAC ONE. All participants will either be contacted by a member of the research team via telephone or ward visit 24 hours (± 4 hours) after BAC ONE dosing to ensure no AEs/SAEs were experienced. The participant's involvement in the study is concluded when the 24 hour assessment has been successfully completed and all AEs/SAEs have been resolved.

ELIGIBILITY:
Inclusion Criteria:

All cohorts

* ≥ 16 years
* Attending consultant permission for bronchoscopy

Cohort 1

* Patients scheduled to undergo surgery under general anaesthesia
* Absence of acute or significant chronic lung disease as determined by the clinical suspicion of the attending medical team or of a medically qualified member of the study investigation team.
* Scheduled presence of an endo-tracheal tube (ETT).
* Capacity to provide informed consent

Cohort 2 and 3

* Patients with bronchiectasis with known microbiological predominance of gram-negative or gram-positive bacteria.
* Capacity to provide informed consent

Cohort 4

* Patients in the ICU with suspected VAP and pulmonary infiltrates on radiological assessment
* Presence of invasive tracheal ventilation tube
* Provision of informed consent from the patient or their personal legal representative prior to any study related procedures.

Exclusion Criteria:

All cohorts

* Refusal for participation by attending consultant
* Any history of anaphylaxis
* Significant coagulopathy, which causes bronchoscopy to be unsuitable, as determined by clinical co-investigator or the participant's attending consultant, using information which is routinely available
* Myocardial infarction in the preceding four weeks
* Women who are pregnant or are breastfeeding
* Receiving drugs that cause increased autofluorescence in the lung, specifically amiodorane and methotrexate

Participants in cohort 4 only

* Inspired Oxygen Concentration (FiO2) >70%
* Positive End Expiratory Pressure (PEEP) >10cm
* ETT or tracheostomy internal diameter < 7mm
* Presence of pneumothorax
* Active bronchospasm
* Mean arterial pressure <65mmHg AND on vasopressor
* Platelet count < 50 x 109/L

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The measurement of BAC ONE fluorescence intensity in the distal lung | Fluorescence signal can be detected within a couple of minutes following BAC ONE administration. On average, signal analysis will be completed within one week of the procedure.
  The main primary outcome measure is to visualise the delivery of BAC ONE in the distal lung of both ventilated controls and patients with acute or chronic bacterial lung infection through the measurement of fluorescence using FE and Cellvizio viewer software.

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MBChB, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No